CLINICAL TRIAL: NCT06516757
Title: A Single Group Study to Evaluate the Effects of a Boric Acid Suppository on Vaginal Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Love Wellness (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20412
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Vaginal Health; Bacterial Vaginosis
Keywords: Vaginal pH Balance; Vaginal Flora; Women's Health
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Boric Acid Suppository Group (Experimental): Participants will use 600 mg Boric Acid Gelatin Capsules (The Killer®) once daily for 7 consecutive days when they feel they are experiencing any signs of vaginal imbalance such as vaginal malodor, irritation, and/or itching.
  Interventions: Dietary Supplement: Boric Acid Suppository

INTERVENTIONS:
Dietary Supplement: Boric Acid Suppository — Participants will complete a baseline questionnaire and a vaginal pH test before using the product, and additional questionnaires and a pH test after 3 and 7 days of product use.
  Other Names: The Killer®

SUMMARY:
This is a virtual single-group clinical trial that will last 12 weeks. Participants will use The Killer® (Boric Acid Suppositories) once daily for 7 consecutive days when they feel that they are experiencing any of the common signs of vaginal imbalance like vaginal malodor, vaginal irritation, and/or vaginal itching. Participants will complete a questionnaire before using the product and on Days 3 and 7 of using the product. They will also complete a vaginal swab pH test before using the product and after 7 days of using the product (Day 8).

ELIGIBILITY:
Inclusion Criteria:

* Female at birth
* Aged 18+
* Interested in maintaining a calm, soothed, and healthy vaginal environment and balanced vaginal pH levels
* Regularly experience atypical vaginal smell, discharge, itching, swelling, irritation, pain or - burning during sex, and/or a burning sensation while urinating
* Willing to avoid introducing any products or new forms of prescription medication or supplements targeting vaginal health during the study period
* Has used a boric acid suppository before
* Willing to avoid the use of any intra-vaginal products during the study product use
* Willing and able to follow the study protocol

Exclusion Criteria:

* Surgeries or invasive treatments in the last six months or planned during the study period
* Introduced any products or forms of prescription medication or supplements targeting vaginal health in the last 12 weeks
* Known allergies to the product ingredients
* Diagnosed with chronic health conditions impacting participation
* Pregnant, breastfeeding, or trying to conceive
* History of substance abuse
* Current or former smoker within the past six months
* Unwilling to follow the study protocol
* Currently participating in any other clinical trial or perception study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Vaginal Health and Balance | Baseline, Day 3, Day 7, and Day 8
  Evaluation of vaginal health and balance via participant questionnaires.
Vaginal Health and Balance | Baseline, and Day 8
  Vaginal pH testing

SECONDARY OUTCOMES:
Participant Perception of Product Convenience | Day 3 and Day 7
  Assessment of participant perception of the convenience of the boric acid suppository compared to other boric acid suppositories via questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No